CLINICAL TRIAL: NCT00884273
Title: A Randomised, Parallel-arm, Open-label Trial Comparing Degarelix With Goserelin Plus Anti-androgen Flare Protection (Bicalutamide), in Terms of Volume Reduction of the Prostate in Patients With Prostate Cancer Being Candidates for Medical Castration
Brief Title: Investigation of the Effect of Degarelix in Terms of Prostate Volume Reduction in Prostate Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS31; 2008-008604-40 (EudraCT Number)
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Degarelix 240 mg/80 mg (Experimental): The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The second and third doses of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections on Days 28 and 56, respectively.
  Interventions: Drug: Degarelix
- Goserelin (3.6 mg) + bicalutamide (50 mg) (Active Comparator): Goserelin implants (3.6 mg) were inserted s.c. into the abdominal wall every 28 days. The first dose was administered on Day 0. The second and third doses of goserelin were administered on Days 28 and 56, respectively.
  On Day 0, participants began once-daily per-oral (p.o.) treatment with bicalutamide (50 mg) as anti-androgen flare protection; this treatment continued for 28 days after the first dose of goserelin.
  Interventions: Drug: Goserelin; Drug: Bicalutamide

INTERVENTIONS:
Drug: Degarelix — The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The second and third doses of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections on Days 28 and 56, respectively.
  Other Names: FE200486; FIRMAGON
  Arms: Degarelix 240 mg/80 mg
Drug: Goserelin — Goserelin implants (3.6 mg) were inserted s.c. into the abdominal wall every 28 days. The first dose was administered on Day 0. The second and third doses of goserelin were administered on Days 28 and 56, respectively.
  Other Names: ZOLADEX
  Arms: Goserelin (3.6 mg) + bicalutamide (50 mg)
Drug: Bicalutamide — On Day 0, participants began once-daily per-oral (p.o.) treatment with bicalutamide (50 mg) as anti-androgen flare protection; this treatment continued for 28 days after the first dose of goserelin.
  Other Names: CASODEX
  Arms: Goserelin (3.6 mg) + bicalutamide (50 mg)

SUMMARY:
This was a Phase 3b clinical study in prostate cancer patients which aimed to compare the current standard therapy of a gonadotrophin releasing hormone (GnRH) agonist, goserelin (3.6 mg; plus anti-androgen flare protection, bicalutamide), to a novel GnRH antagonist, degarelix (240 mg starting dose/80 mg maintenance dose) with respect to mean percentage reduction in prostate volume.

The hypothesis was that degarelix could decrease prostate size at least as effectively as the combination of a GnRH agonist with an anti-androgen for flare protection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has given written informed consent
2. Patient is 18 years or older
3. Patient has histologically confirmed prostate cancer
4. Patient has a serum prostate-specific antigen (PSA) level at screening >2 ng/mL
5. The prostate size is >30 cubic centimetres (cc), measured by TRUS
6. Patient has had a bone-scan within 12 weeks before inclusion
7. Patient must be able to undergo transrectal examinations
8. Patient has an estimated life expectancy of at least 12 months

Exclusion Criteria:

1. Any previous treatments for prostate cancer
2. Previous trans-urethral resection of the prostate (TURP)
3. Is not considered a candidate for medical castration
4. Use of urethral catheter
5. Is currently treated with a 5-alpha reductase inhibitor
6. Is currently treated with an alpha-adrenoceptor antagonist
7. Treatment with botulinum toxin A (Botox)
8. Require radiotherapy during the trial
9. History of severe untreated asthma, anaphylactic reactions, or severe urticaria and/or angioedema
10. Hypersensitivity towards any component of the investigational products or excipients
11. Previous history or presence of another malignancy
12. A clinically significant disorder
13. A corrected QT interval over 450 msec
14. Mental incapacity or language barrier precluding adequate understanding or co-operation
15. Receipt of an investigational drug within the last 28 days proceeding screening
16. Previous participation in any degarelix trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (46):
- Belgium (4):
  - Hospital St Jan Brugge, Bruges
  - Institut Jules Bordet, Brussels
  - University Hospitals Leuven, Leuven
  - St. Elisabethziekenhuis, Turnhout
- Denmark (6):
  - Aalborg Sygehus syd, Aalborg
  - Århus Universitetshospital, Skejby, Aarhus
  - Herlev Hospital, Ballerup Municipality
  - Regionhospitalet Holstebro, Holstebro
  - Sygehus Syd, Næstved Sygehus, Næstved
  - Roskilde Sygehus, Roskilde
- Finland (4):
  - HYKS/kirurgian klin./urologia, Helsinki
  - KYS/kirurgian klin (Kuopio), Kuopio
  - OYS/kirurgian klinik, Oulu
  - TAYS/kirurgian klinik, Tampere
- Italy (13):
  - Azienda Ospedaliero Universitaria Ospedali riuniti, Ancona
  - Azienda Ospedaliera S. Giuseppe Moscaaati, Avellino
  - Policlinico S.Orsola Malpighi - Universita' degli Studi di Bologna, Bologna
  - U.O. Di Urologia - Spedali Civili di Brescia, Brescia
  - Clinica Urologica 1 Universita. Firensa, Florence
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Fondazione IRCCS Ospedale Maggiore Policlinico Mangiagalli e Regina Elena, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone dell'Universita' degli Studi di Palermo, Palermo
  - Clinica Urologica - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliera S. Andrea - Universita' la Sapienza di Roma, Roma
  - S.C. Di Urologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliero Universitaria S. Giovanni Battista - Molinette, Torino
- Norway (4):
  - Moelv spesialistsenter, Moelv
  - Aker Universitetssykehus HF, Oslo
  - Det Norske Radiumhospitalet HF, Oslo
  - St Olavs Hospital HF, Trondheim
- Portugal (4):
  - Hospital Fernando da Fonseca, Amadora
  - Hospitais Universidade Coimbra, Coimbra
  - Centro Hospitalar Lisboa Norte, Hospital Santa Maria, Lisbon
  - Hospital S.João, Porto
- Sweden (6):
  - Investigational site, Gothenburg
  - SU/Sahlgrenska, Gothenburg
  - Helsingborgs Lasarett, Helsingborg
  - Universitetssjukhuset MAS, Malmo
  - Södertälje Sjukhus, Södertälje
  - Uppsala/Akademiska sjukhuset, Uppsala
- Turkey (Türkiye) (5):
  - Cerrahpasa Faculty of Medicine, Kocamustafapasa, Istanbul
  - Istanbul University Faculty of Medicine, ÇAPA, Istanbul
  - Marmara University Faculty of Medicine, Altunizade, Istanbul
  - Ankara University Faculty of Medicine, Sıhhıye - Ankara
  - Hacettepe University Faculty of Medicine, Sıhhıye - Ankara

REFERENCES:
- [Result] Axcrona K, Aaltomaa S, da Silva CM, Ozen H, Damber JE, Tanko LB, Colli E, Klarskov P. Androgen deprivation therapy for volume reduction, lower urinary tract symptom relief and quality of life improvement in patients with prostate cancer: degarelix vs goserelin plus bicalutamide. BJU Int. 2012 Dec;110(11):1721-8. doi: 10.1111/j.1464-410X.2012.11107.x. Epub 2012 Apr 13. PMID 22500884
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited by outpatient urologists. 180 participants were to be randomised in a 1:1 ratio to one of two treatment groups (90 participants were to be treated with degarelix; 90 participants were to be treated with goserelin plus bicalutamide). The recruitment period was August 2009 - December 2010.
Pre-assignment Details: The apparent skewed number of actual participants in the two groups is due to the fact that randomisation was done in blocks per site rather than per study.
Period: Overall Study
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Started | 84 (Intention-to-treat (ITT) population.) | 98 (ITT population.)
Full Analysis Set (FAS) | 82 (Two participants did not have any post-dose efficacy assessment and were excluded from the FAS.) | 97 (One participant did not have any post-dose efficacy assessment and was excluded from the FAS.)
Per Protocol (PP) Analysis Set | 81 | 92
Safety Analysis Set | 84 | 98
Completed | 82 | 93
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — Practical reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg) | Total
Number analyzed (Participants) | 82 | 97 | 179
Age Continuous [Mean (Standard Deviation); unit: years] — Full Analysis Set (FAS).
  years | 71.9 (7.71) | 73.0 (7.10) | 72.5 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants] — FAS.
  Participants
    Female | 0 | 0 | 0
    Male | 82 | 97 | 179
Race (NIH/OMB) [Count of Participants; unit: Participants] — FAS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 82 | 97 | 179
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — FAS.
  participants
    Portugal | 4 | 7 | 11
    Finland | 14 | 17 | 31
    Belgium | 2 | 2 | 4
    Turkey | 14 | 14 | 28
    Denmark | 13 | 15 | 28
    Norway | 4 | 8 | 12
    Italy | 20 | 22 | 42
    Sweden | 11 | 12 | 23
Body Weight [Mean (Standard Deviation); unit: kilogram] — FAS.
  kilogram | 79.7 (12.4) | 79.7 (12.2) | 79.7 (12.2)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] — FAS.
  kilogram per square meter | 26.8 (4.07) | 26.5 (3.72) | 26.6 (3.88)
Gleason Score [Number; unit: participants] — FAS. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    Gleason Score 2-4 | 1 | 1 | 2
    Gleason Score 5-6 | 16 | 15 | 31
    Gleason Score 7-10 | 65 | 81 | 146
Stage of Prostate Cancer [Number; unit: participants] — FAS. Prostate cancer stage was classified according to the Tumor, Nodes, and Metastatic (TNM) scale to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor. Some participants did not have their prostate cancer classified for the complete TNM scale (17 participants).
  participants
    Localized | 24 | 32 | 56
    Locally Advanced | 30 | 23 | 53
    Metastatic | 22 | 31 | 53
    Not Classifiable | 6 | 11 | 17
Serum Testosterone Levels [Median (Full Range); unit: nanograms per milliliter] | 4.08 [0.32 to 10.8] | 4.33 [0.13 to 9.6] | 4.23 [0.13 to 10.8]
Serum Protsate-Specific Antigen (PSA) Levels [Median (Full Range); unit: nanograms per milliliter] | 27.8 [1.9 to 6206] | 15.6 [3.0 to 2829] | 20.2 [1.9 to 6206]
Prostate Volume [Mean (Standard Deviation); unit: milliliter] — Prostate volume was measured with a Trans Rectal Ultrasound Scan (TRUS).
  milliliter | 54.8 (26.0) | 49.9 (15.5) | 52.1 (21.1)
Total International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: scores on a scale] — The IPSS is a tool commonly used to assess the severity of lower urinary tract symptoms (LUTS), and to monitor the progress of the disease once treatment has been initiated. The participant completes a questionnaire containing 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Each question is assigned a score of 0-5. The total score is then classified according to the following scale: 0 to 7 = mildly symptomatic; 8 to 19 = moderately symptomatic; and 20 to 35 = severely symptomatic.
  scores on a scale | 14.3 (6.91) | 13.4 (7.36) | 13.8 (7.15)
Quality of Life (QoL) Related to Urinary Symptoms [Mean (Standard Deviation); unit: scores on a scale] — The IPSS questionnaire included an additional single question to assess the participant's QoL in relation to his urinary symptoms. The question was: 'If you were to spend the rest of your life with your urinary condition the way it is now, how would you feel about that?' The possible answers to this question ranged from 'delighted' (a score of '0') to 'terrible' (a score of '6'). The figures in the tables present the change (ie decrease) in IPSS QoL score, i.e. the bigger the decrease the better QoL.
  scores on a scale | 2.85 (1.62) | 2.73 (1.66) | 2.79 (1.64)
Benign Prostatic Hyperplasia Impact Index (BPHII) [Mean (Standard Deviation); unit: scores on a scale] — The Benign Prostatic Hyperplasia Impact Index (BPHII) is a self-administered questionnaire to measure how much urinary problems affect various domains of health. The higher value the worse are the urinary problems. The minimum possible total value is 0 and the maximum possible total value is 16.
  scores on a scale | 5.06 (3.39) | 4.58 (3.58) | 4.80 (3.49)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Prostate Size Based on Trans Rectal Ultra Sound (TRUS) at Week 12 (Full Analysis Set)
Description: TRUS is a method of measuring the size of the prostate.
Time Frame: After treatment of 12 weeks compared to Baseline
Population: Full Analysis Set (FAS), Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 82 | 97
milliliter | -37.2 (16.8) | -39.0 (17.7)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); Estimates from analysis of variance with treatment as factors and baseline IPSS and baseline Prostate volume as covariates; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be established if the treatment difference in adjusted (for baseline volume, and baseline total IPSS) mean percentage reduction was significantly greater (two-sided at α=0.05 level) than Δ = 10 points (non-inferiority margin) in both the FAS and PP analyses sets. If the Week 12 treatment assessment of prostate volume was missing the LOCF approach was used, i.e., the prostate volume value closest to and before Week 12 was used; p = 0.36, ANCOVA — FAS; The baseline IPSS and baseline Prostate volume were used as covariates and treatment was used as a factor in the analysis; Mean Difference (Final Values) = 2.37, 95% CI 2-sided [-2.78 to 7.52]

2. Secondary Outcome: Change From Baseline in Prostate Size Based on TRUS at Week 4 and 8
Description: TRUS is a method of measuring the size of the prostate.
Time Frame: After treatment of 4 and 8 weeks compared to Baseline
Population: FAS, Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 82 | 97
milliliter
  Week 4 | -19.2 (15.2) | -21.2 (17.7)
  Week 8 | -33.1 (14.8) | -33.2 (20.6)

3. Secondary Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS) at Week 4, 8, and 12
Description: The IPSS is a tool commonly used to assess the severity of lower urinary tract symptoms (LUTS), and to monitor the progress of the disease once treatment has been initiated. The participant completes a questionnaire containing 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Each question is assigned a score of 0-5. The total score is then classified according to the following scale: 0 to 7 = mildly symptomatic; 8 to 19 = moderately symptomatic; and 20 to 35 = severely symptomatic.
Time Frame: After treatment of 4, 8, and 12 weeks compared to Baseline
Population: FAS, Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 82 | 97
scores on a scale
  Week 4 | -2.09 (4.36) | -1.36 (5.86)
  Week 8 | -3.55 (5.95) | -3.13 (6.06)
  Week 12 | -4.39 (6.66) | -2.74 (6.37)

4. Secondary Outcome: Change in Serum Testosterone Levels During the Study
Time Frame: At 4, 8, and 12 weeks compared to baseline.
Population: FAS.
Measure: Median (Full Range); unit: nanograms per milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 82 | 97
nanograms per milliliter
  Week 4 | -3.91 [-10.62 to -0.20] | -4.17 [-9.30 to 0.03]
  Week 8 | -3.97 [-10.61 to -0.12] | -4.24 [-9.44 to -0.08]
  Week 12 | -4.09 [-10.58 to 0.00] | -4.23 [-9.31 to -0.03]

5. Secondary Outcome: Change in Serum Prostate-Specific Antigen (PSA) Levels During the Study
Time Frame: At 4, 8, and 12 weeks compared to baseline.
Population: FAS.
Measure: Median (Full Range); unit: nanograms per milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 82 | 97
nanograms per milliliter
  Week 4 | -20.25 [-4205 to 4.5] | -12.10 [-2823 to 3.3]
  Week 8 | -22.5 [-6192 to 4.3] | -14.6 [-2828 to -2]
  Week 12 | -25.15 [-6195 to 4.7] | -13.1 [-2815 to -1.2]

6. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Related to Urinary Symptoms at Each Visit
Description: The IPSS questionnaire included an additional single question to assess the participant's QoL in relation to his urinary symptoms. The question was: 'If you were to spend the rest of your life with your urinary condition the way it is now, how would you feel about that?' The possible answers to this question ranged from 'delighted' (a score of '0') to 'terrible' (a score of '6').
Time Frame: After treatment of 4, 8, and 12 weeks compared to Baseline
Population: FAS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 82 | 97
scores on a scale
  Week 4 | -0.46 (1.43) | -0.56 (1.30)
  Week 8 | -0.83 (1.62) | -0.79 (1.37)
  Week 12 | -0.99 (1.64) | -1.01 (1.38)

7. Secondary Outcome: Change From Baseline in Burden of Urinary Symptoms Based on the Benign Prostatic Hyperplasia Impact Index (BPHII)
Description: The Benign Prostatic Hyperplasia Impact Index (BPHII) is a self-administered questionnaire to measure how much urinary problems affect various domains of health. The higher value the worse are the urinary problems. The minimum possible total value is 0 and the maximum possible total value is 16.
Time Frame: After treatment of 4, 8, and 12 weeks compared to Baseline
Population: FAS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 82 | 97
scores on a scale
  Week 4 | -0.78 (2.03) | -0.70 (2.34)
  Week 8 | -0.88 (2.73) | -1.09 (2.48)
  Week 12 | -1.28 (2.62) | -1.16 (2.67)

8. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The table presents the number of participants with normal baseline and at least one post-baseline markedly abnormal value.
Time Frame: Baseline to 12 weeks of treatment
Population: Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 84 | 98
participants
  Diastolic blood pressure <=50 and decrease >=15 | 0 | 0
  Diastolic blood pressure >=105 and increase >=15 | 0 | 1
  Systolic blood pressure <=90 and decrease >=20 | 0 | 0
  Systolic blood pressure >=180 and increase >=20 | 2 | 4
  Heart rate <=50 and decrease >=15 | 1 | 0
  Heart rate >=120 and increase >=15 | 0 | 0
  Body weight decrease of >=7 percent | 0 | 5
  Body weight increase of >=7 percent | 2 | 3

9. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Safety Laboratory Variables
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) levels of safety laboratory variables. Only the laboratory variables that had at least one percentage of participants in either group with abnormal value are presented, more variables were included in the study.
Time Frame: Baseline to 12 weeks of treatment
Population: Safety Analysis Set.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 84 | 98
participants
  B-Haematocrit (Ratio) <=0.37 | 13 | 16
  B-Haemoglobin (g/L) <=115 | 2 | 1
  B-Red blood cell count (10^12/L) <=3.5 | 1 | 0
  B-White blood cell count (10^9/L) <=2.8 | 3 | 1
  S-Alanine aminotransferase (IU/L) >3xULN | 1 | 2
  S-Alkaline phosphatase (IU/L) >3xULN+25% increase | 0 | 1
  S-Aspartate aminotransferase (IU/L) >3xULN | 0 | 2
  S-Cholesterol (mmol/L) >=8.0 | 2 | 0
  S-Glutamyltransferase (IU/L) >3xULN | 1 | 0
  S-Potassium (mmol/L) >=5.8 | 3 | 3
  S-Urea nitrogen (mmol/L) >=10.7 | 10 | 3

10. Primary Outcome: Change From Baseline in Prostate Size Based on Trans Rectal Ultra Sound (TRUS) at Week 12 (Per Protocol Analysis Set)
Description: TRUS is a method of measuring the size of the prostate.
Time Frame: After treatment of 12 weeks compared to Baseline
Population: Per Protocol (PP) Analysis Set, Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 81 | 92
milliliter | -37.3 (16.8) | -39.0 (18.4)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.41, ANCOVA — PP; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 2.24, 95% CI 2-sided [-3.10 to 7.58]

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Serious Adverse Events (participants affected / at risk) | 1/84 | 7/98
Other Adverse Events (participants affected / at risk) | 33/84 | 47/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/80 mg (N=84) | Goserelin (3.6 mg) + Bicalutamide (50 mg) (N=98)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter related complication (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/80 mg (N=84) | Goserelin (3.6 mg) + Bicalutamide (50 mg) (N=98)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 12 (20) | 0 (0)
Injection site erythema (General disorders) | 3 (4) | 0 (0)
Injection site swelling (General disorders) | 3 (4) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Injection site induration (General disorders) | 2 (4) | 0 (0)
Injection site inflammation (General disorders) | 2 (2) | 0 (0)
Injection site pruritus (General disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 4 (5) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Hot flush (Vascular disorders) | 8 (8) | 17 (17)
Flushing (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.